CLINICAL TRIAL: NCT03748511
Title: Identification of Microbial Properties Predicting a Worsening Course of Fatty Liver Disease
Acronym: FLM
Status: Terminated | Type: Observational
Why Stopped: COVID-19 interrupted the recruitment process and imposed difficulties
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Rawi Hazzan, Head of Liver Unit, HaEmek Medical Center, Israel
Other Study IDs: 179-17-EMC
Record Dates: First submitted 2018-09-17; First posted 2018-11-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Patients With Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- fatty liver disease 0-1F: 20 patients with uncomplicated liver disease, with fibrosis stage 0-1F.
  Interventions: Other: fibroscan and stool sample
- fatty liver disease 2F: 20 patients with liver disease, fibrosis stage 2F.
  Interventions: Other: fibroscan and stool sample
- fatty liver disease 3-4F: 20 patients with advanced liver disease, fibrosis stage 3-4F.
  Interventions: Other: fibroscan and stool sample

INTERVENTIONS:
Other: fibroscan and stool sample — patients undergo ultrasaound (fibroscan) in order to stage the liver disease.
  Other Names: fibroscan is also called shear wave

SUMMARY:
This study investigates the relation between the gastrointestinal tract bacteria and the progression of fatty liver disease .

DETAILED DESCRIPTION:
In the gastrointestinal (GI) tract live wide spectrum of bacteria, in this study we are trying to find if there is a relation between the GI tract bacteria and the development of non alcoholic fatty liver disease, the results of the this study may help us identify the stage of liver disease in noninvasive means and enables us to adopt methods to reduce morbodity.

ELIGIBILITY:
Inclusion Criteria:

* patients with non alcoholic fatty liver disese.
* patients who give approval to participate in the study

Exclusion Criteria:

* liver failure
* acute or chronic kidney failure
* heart failure ( NYHA 3-4)
* active cancer
* fatty liver due to non alcoholic etiology.
* patients who consume drugs from the estrogen/methotrexate family, or chloroquine.
* history of hypothyrodism or cushing.
* patients who used TPA in the last 6 months .
* pathients with chronic liver disease like A1AT, hemochromatosis, wilson, toxic damage and autoimmunity .
* special population like - children, pregnant women and patients who lack the ability to make judgment.
* infectious liver disease - viral hepatitis or HIV.
* inflammatory bowel disease.
* patients who underwent surgery of the gastrointestinal trant.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 patients with fatty liver disease
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Transient Elastography Test | up to 2 hours
  Ultrasound Elastography is a non-invasive test which uses the technology of Shear Wave Elastography (SWE) obtained from the right liver lobe for staging liver fibrosis according to Metavir Fibrosis Score .
  Metavir Fibrosis Score is a system used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy.
  Liver fibrosis assessed by Shear Wave Elastography is well correlated to biopsy using Metavir Score.
  The outcome of the test will be correlated to Metavir Score system according to the chart below:
  SWE (kiloPascal) , METAVIR score, Fibrosis Level. Below 5 , F0 , No fibrosis. 5.0-7.1 , F1 , Mild Fibrosis. 7.1-8.7 , F2 , Significant Fibrosis. 8.7-10.4 , F3 , Sever Fibrosis . 10.4-19 , F4 , Cirrhosis.

SECONDARY OUTCOMES:
Gastrointestinal Microbiome test | up to 1 month
  The test will be made by a new meta-genomic sequencing technology (Next Generation Sequencing) which gives us unbiased information about all the gastrointestinal bacterial characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Init, Afula, Israel

IPD SHARING:
Plan to Share IPD: No